CLINICAL TRIAL: NCT07042438
Title: A Phase 2 Randomized Trial of Remodeling Intestinal Microbiota Using Fecal Microbiome Transplant (FMT) Among Recipients of Chimeric Antigen Receptor T Cells (CAR T)
Brief Title: Fecal Microbiome Transplant to Remodel Intestinal Microbiota for Patients With Relapsed or Refractory Lymphoma With Exposure to High-Risk Antibiotics Who Are Receiving Chimeric Antigen Receptor T Cells
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24910; NCI-2025-03771 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24910 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-06-06; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Recurrent Diffuse Large B-Cell Lymphoma; Recurrent High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; Recurrent Transformed Follicular Lymphoma to Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; Refractory Transformed Follicular Lymphoma to Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — axicabtagene ciloleucel; Specimen Handling; Drug Therapy; Fecal Microbiota Transplantation; Leukapheresis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This single center, double-blind, phase 2a clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (FMT) (Experimental): Patients undergo standard of care leukapheresis and receive standard of care chemotherapy and CAR T cells. Patients receive FMT PO QD on day -10 and -7 before leukapheresis, day -10 and -7 before CAR T cell infusion, within 3 days of neutrophil recovery and 2 days after first neutrophil recovery dose. Treatment given in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study.
  Interventions: Biological: Axicabtagene Ciloleucel; Procedure: Biospecimen Collection; Drug: Chemotherapy; Procedure: Fecal Microbiota Transplantation; Procedure: Leukapheresis
- Arm II (Placebo) (Placebo Comparator): Patients undergo standard of care leukapheresis and receive standard of care chemotherapy and CAR T cells. Patients receive placebo PO QD on day -10 and -7 before leukapheresis, day -10 and -7 before CAR T cell infusion, within 3 days of neutrophil recovery and 2 days after first neutrophil recovery dose. Treatment given in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Chemotherapy; Procedure: Fecal Microbiota Transplantation; Procedure: Leukapheresis; Drug: Placebo Administration

INTERVENTIONS:
Biological: Axicabtagene Ciloleucel — Given CAR-T cells
  Other Names: Axi-cel; Axicel; KTE C19; KTE-C19; KTE-C19 CAR; KTEC19; Yescarta
  Arms: Arm I (FMT)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Chemotherapy — Receive chemotherapy
  Other Names: Chemo; Chemotherapy (NOS); Chemotherapy, Cancer, General
Procedure: Fecal Microbiota Transplantation — Given PO
  Other Names: Fecal Material Transplantation; Fecal Transplantation; FMT; Poo Transplant; Poop Transplant; Stool Transplant
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocyte Adsorptive Apheresis; Leukocytopheresis; Therapeutic Leukopheresis; White Blood Cell Reduction Apheresis
Drug: Placebo Administration — Given PO
  Arms: Arm II (Placebo)

SUMMARY:
This phase II trial tests how well fecal microbiome transplantation works to remodel intestinal microbiota for patients with lymphoma that has come back after a period of improvement (relapsed) or that does not respond to treatment (refractory) with exposure to high-risk antibiotics who are receiving chimeric antigen receptor (CAR) T cells. Fecal microbiome transplantation consists of fecal microbiota from healthy donors with healthy gut microbiota that allows re-population of the patient's microbiome with diverse protective microorganisms. CAR T-cell therapy is a type of treatment in which a patient's T cells (a type of immune system cell) are changed in the laboratory so they will attack cancer cells. T cells are taken from a patient's blood. Then the gene for a special receptor that binds to a certain protein on the patient's cancer cells is added to the T cells in the laboratory. The special receptor is called a chimeric antigen receptor (CAR). Large numbers of the CAR T cells are grown in the laboratory and given to the patient by infusion for treatment of certain cancers. Part of the treatment for CAR T therapy involves high doses of chemotherapy. This, along with prior exposure to high strength antibiotics, can damage patient's intestinal microbiota. Giving fecal microbiome transplantation may improve clinical response by repairing intestinal microbiota for patients with relapsed or refractory lymphoma who had exposure to high-risk antibiotics.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the efficacy of fecal microbiome transplant (FMT) by measuring changes in gut microbiome diversity (as assessed by Shannon alpha diversity Index) at day 0 (day of CAR T infusion).

SECONDARY OBJECTIVES:

I. Estimate rates of complete response (CR) at days +30, +90 or 1 year after CAR T therapy in each arm. (Key secondary objective) II. Determine the safety and tolerability/feasibility of fecal microbiota transplant (FMT) until 28 days post last dose by adverse events: type, frequency, severity, attribution, time course, duration.

III. Quantify engraftment of bacterial strains that are definitely attributable to FMT product.

IV. Estimate incidence and severity of cytokine release syndrome (CRS) and immune effector cell associated neurotoxicity syndrome (ICANS) in each arm.

V. Shannon index at each fecal sampling timepoint after day 0 to assess overtime changes in microbiome diversity in each cohort after CAR T infusion.

VII. Estimate rates of overall response (ORR) at 30 days, 90 days and 1 year after CAR T therapy in each arm.

VIII. Determine the number of bacterial infection rate post 30 days of last FMT last dose.

IX. Estimate rate of overall survival (OS), relapse/progression and non-relapse mortality (NRM) at 30 days, 90 days and 1 year after CAR T therapy in each arm.

X. Estimate time to neutropenia recovery at each arm.

EXPLORATORY OBJECTIVES:

I. Compare quality of manufactured CAR T products in patients treated or not treated with FMT.

II. Characterize and correlate FMT treatment with the following biologic endpoints.

IIa. Plasma and stool metabolites with a focus on butyrate-related pathways (metabolomics analysis); IIb. T cell phenotype (multicolor flow cytometry at Immuno-Oncology Core) and cytokines assay (30-multiplex plate using Luminex); IIc. CAR T cell persistence (using standard polymerase chain reaction [PCR] assays) on days +30, +90, 6 months and 1 year after CAR T therapy.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo standard of care leukapheresis and receive standard of care chemotherapy and CAR T cells. Patients receive FMT orally (PO) once daily (QD) on day -10 and -7 before leukapheresis, day -10 and -7 before CAR T cell infusion, within 3 days of neutrophil recovery and 2 days after first neutrophil recovery dose. Treatment given in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study.

ARM II: Patients undergo standard of care leukapheresis and receive standard of care chemotherapy and CAR T cells. Patients receive placebo PO QD on day -10 and -7 before leukapheresis, day -10 and -7 before CAR T cell infusion, within 3 days of neutrophil recovery and 2 days after first neutrophil recovery dose. Treatment given in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study.

After completion of study treatment, patients are followed up at day 28, 90 and 1 year post CAR T cell therapy.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative.

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Age: ≥ 18 years
* Karnofsky performance status (KPS) ≥ 60
* Confirmed diagnosis of relapsed/refractory CD19 B-cell lymphomas of diffuse large B cell lymphoma (DLBCL), transformed follicular lymphoma (tFL), or double-hit lymphoma (DHL) and scheduled to receive commercial CAR T treatment of YESCARTA ® for their diagnosis
* Fully recovered from the acute toxic effects (except alopecia) to ≤ grade 1 to prior anti-cancer therapy
* Exposure to high-risk antibiotics within 90 days of consent. High-risk broad-spectrum antibiotics include carbapenems (meropenem, imipenem, doripenem), anti-pseudomonal antibiotics (cefepime, piperacillin-tazobactam, ceftazidime) or anaerobic antibiotics including metronidazole, clindamycin, amoxicillin-sulbactam, and vancomycin
* Clinical laboratory and organ function criteria per standard of care to CAR T patients at City of hope: (To be performed within 30 days prior to leukapheresis)
* Seronegative for HIV antigen (Ag)/antibody (Ab) combo, hepatitis C virus (HCV), active hepatitis B virus (HBV) (surface antigen negative)

  * HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* Meets other institutional and federal requirements for infectious disease titer requirements

  * Note: Infectious disease testing to be performed within 28 days prior to day 1 of protocol therapy
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential* to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 12 months after the last dose of protocol therapy.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Major surgery in 4 months preceding enrollment
* No live vaccine in 30 days prior to enrollment
* Inability to swallow capsules or history of disorder with Inability to swallow FMT capsules
* History of inflammatory bowel disorder, irritable bowel disorder
* Severe food allergies
* History of chronic aspiration
* History of behavioral disorders including substance abuse disorders which per discretion of primary investigator will interfere with safe conduct and compliance to study treatment
* History neurocognitive disorder which per discretion of primary investigator will interfere with safe conduct and compliance to study treatment
* Diagnosis of primary immunodeficiency
* Active second malignancy requiring treatment except non-melanoma skin cancer or carcinoma in situ-cervix, bladder or to non-metastatic prostate cancer which does not require treatment
* Uncontrolled bacterial, fungal, or viral infection confirmed using clinical, laboratory and radiological findings requiring administration of intravenously (IV) antimicrobials
* Any clinical, laboratory or radiologic findings per discretion of primary investigator will interfere with safe conduct of study treatment and compliance with study procedures
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-01-17 (Estimated); Primary Completion 2028-04-13 (Estimated); Study Completion 2028-04-13 (Estimated)

PRIMARY OUTCOMES:
Changes in gut microbiome diversity | From baseline to day 0
  Assessed using the Shannon alpha diversity index. For comparisons at a timepoint of most interest, a t-test (or Wilcoxon rank-sum test if assumptions are not met) will be used to compare the Shannon index between the fecal microbiome transplant (FMT) and placebo groups. For over-time comparisons, linear mixed models will be used to assess longitudinal changes in microbiome diversity between treatment (FMT) and control (placebo) groups, accounting for within-subject correlations over multiple measurement points.

SECONDARY OUTCOMES:
Rate of complete response | At day +30, +90 and 1 year after chimeric antigen receptor t cell (CAR T) therapy
Incidence of adverse events | Up to 1 year post CAR T cell therapy
  Scored using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 scale. Will summarize adverse events by type, severity, attribution, time of onset, duration, and association with study treatment. All observed toxicities will be tabulated and summarized by grade and frequency.
Feasibility of Rx administration | Up to 30 days before CAR T cell infusion
  Evaluated by assessment of patient's ability to take at least 2 of the first 4 doses of Rx (4 capsules of FMT or placebo) before CAR T infusion.
Quantify engraftment of bacterial strains that are definitely attributable to FMT product | Up to 1 year post CAR T cell therapy
  Donor microbiota engraftment will be determined by SourceTracker. SourceTracker estimates the attribution of microbiota in a post-treatment sample to donor microbiota. In choosing the donor source for each post-FMT sample, only the specific donor whose product was administered to the patient was used as donor. By contrast, because placebo capsules did not contain any donor material, the calculated engraftment rates from all four presumptive donors were averaged to derive donor attribution of post-placebo microbiota.
Incidence and severity of Cytokine Release Syndrome | Up to 1 year post CAR T cell therapy
Incidence and severity of immune effector cell associated neurotoxicity syndrome | Up to 1 year post CAR T cell therapy
Overall response rate | At day +30, +90 and 1 year after CAR T therapy
  The binomial exact 95% confidence interval will be estimated at each post-treatment assessment timepoint and compared between FMT and placebo by Pearson Chi-square test or Fisher exact test.
Bacterial infection rate | Post 30 days of last FMT last dose
Rate of overall survival | At day +30, +90 and 1 year after CAR T therapy
Rate of relapse/progression | At day +30, +90 and 1 year after CAR T therapy
Rate of non-relapse mortality | At day +30, +90 and 1 year after CAR T therapy
  The binomial exact 95% confidence interval will be estimated at each post-treatment assessment timepoint and compared between FMT and placebo by Pearson Chi-square test or Fisher exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Karamjeet S Sandhu, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States